CLINICAL TRIAL: NCT01607853
Title: A Phase IIa Exploratory Study Evaluating the Anti-psoriatic Effect of Daivobet® Gel Applied Then Removed After 10 Minutes, Daivobet® Gel Applied Then Removed After 20 Minutes, Daivobet® Gel Applied for 24 Hours and Daivobet® Gel Vehicle Applied for 24 Hours
Brief Title: A Short-contact Plaque Test Study With Daivobet® Gel in Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: LP0076-57; 2012-001507-21 (EudraCT Number)
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daivobet® gel (Experimental)
  Interventions: Drug: Daivobet® gel applied then removed after 10 minutes (+/- 2 minutes); Drug: Daivobet® gel applied then removed after 20 minutes (+/- 2 minutes); Drug: Daivobet® gel applied for 24 hours (+/- 2 hours); Drug: Daivobet® gel vehicle applied for 24 hours (+/- 2 hours)

INTERVENTIONS:
Drug: Daivobet® gel applied then removed after 10 minutes (+/- 2 minutes) — Once daily application, 3 weeks
Drug: Daivobet® gel applied then removed after 20 minutes (+/- 2 minutes) — Once daily application, 3 weeks
Drug: Daivobet® gel applied for 24 hours (+/- 2 hours) — Once daily application, 3 weeks
Drug: Daivobet® gel vehicle applied for 24 hours (+/- 2 hours) — Once daily application, 3 weeks

SUMMARY:
The purpose of this study is to evaluate the anti-psoriatic effect of Daivobet® gel applied then removed after 10 minutes (+/- 2 minutes), Daivobet® gel applied then removed after 20 minutes (+/- 2 minutes) compared with Daivobet® gel and Daivobet® gel vehicle applied for 24 hours (+/- 2 hours), using the psoriasis plaque test modified from the method developed by KJ Dumas and JR Scholtz.

ELIGIBILITY:
Inclusion Criteria:

1. Following verbal and written information about the trial, the subject has to provide signed and dated informed consent before any study related activities are carried out.
2. Age 18 years or above.
3. Either sex.
4. All skin types.
5. Subjects with a diagnosis of psoriasis vulgaris with lesions located on arms, legs and/or trunk. The lesions must have a total size suitable for application of 4 different products.
6. Subjects with, in the opinion of the investigator, stable psoriasis based on Total Plaque Score evaluated at screening visit and at visit 2 (baseline).
7. Subjects with psoriasis lesions (plaques) assessed by a Total Clinical Score (sum of scores of erythema, scaling and infiltration) of 4 to 9 inclusive, but each individual item ≥ 1.
8. Subjects willing and able to follow all the study procedures and complete the whole study.
9. Subjects affiliated to a social security system.
10. Female subjects of childbearing potential using a reliable method of contraception for at least 1 month before the study start and during the course of the study (e.g., oral contraceptive pill, intrauterine device, contraceptive patches, implantable contraception, condoms) or females of non-childbearing potential (i.e. postmenopausal (absence of menstrual bleeding for 2 years), hysterectomy, bilateral ovariectomy or tubal section/ligation).
11. Female with a negative urine pregnancy test (at screening visit).

Exclusion Criteria:

1. Females who are pregnant, of child-bearing potential and who wish to become pregnant during the study, or who are breast feeding.
2. Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis vulgaris within 4 weeks (etanercept), 2 months (adalimumab, alefacept, infliximab), 4 months (ustekinumab) or 4 weeks/5 half-lives (which-ever is longer) for experimental biological products prior to randomisation and during the study.
3. Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within the 4- week period prior to randomisation and during the study.
4. Use of phototherapy within the following time periods prior to randomisation and during the study:

   * PUVA or Grenz ray therapy (4 weeks),
   * UVB (2 weeks).
5. Subjects using one of the following topical drugs within 4 weeks prior to randomisation and during the study:

   - Potent or very potent (WHO group III-IV) corticosteroids.
6. Subjects using one of the following topical drugs for the treatment of psoriasis within 2 weeks prior to randomisation and during the study:

   * WHO group I-II corticosteroids (except if used for treatment of scalp and/or facial psoriasis),
   * Topical retinoids,
   * Vitamin D analogues,
   * Topical immunomodulators (e.g. calcineurin inhibitors),
   * Anthracen derivatives,
   * Tar,
   * Salicylic acid.
7. Subjects using emollients on the target plaques within one week before randomisation and during the study.
8. Initiation of, or expected changes in concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium and ACE inhibitors) within 2 weeks prior to randomisation and during the study.
9. Subjects with current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis.
10. Subjects with known/suspected disorders of calcium metabolism associated with hypercalcemia within the last 10 years, based on medical history.
11. Subjects with any of the following conditions present on the test area: viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections and atrophic skin.
12. Subjects with skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, icthyosis, acne rosacea, ulcers and wounds within the plaque test areas.
13. History of any severe disease or serious current condition (based on subject interview and/or results of screening physical examination) which, in the opinion of the investigator, would put the subject at risk by participating in the study or would interfere significantly with the evaluation of study results or the study course (e.g. cancer, severe cardiopathy, severe renal insufficiency, severe hepatic insufficiency).
14. Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the 4 week period prior to randomisation or longer, if the class of the substance requires a longer washout as defined above (e.g., biological treatments).
15. Subjects with current participation in any other interventional clinical trial, based on interview of the subject.
16. Subjects with known or suspected hypersensitivity to component(s) of the investigational products.
17. Subjects with any concomitant medical or dermatological disorder(s) which might preclude accurate evaluation of the psoriasis.
18. Subjects foreseeing an intensive solar exposure during the study (UV radiation, etc.) or having been exposed within two weeks preceding the screening visit.
19. Subjects impossible to contact in case of emergency.
20. Subjects who are known or, in the opinion of the investigator, are unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency or psychotic state).
21. Subjects who are in an exclusion period in the National Biomedical Research Register of the French Ministry of Health at randomisation.
22. Subjects under guardianship, hospitalized in a public or private institution, for a reason other than the research or subject deprived of freedom.
23. Subjects previously randomised in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, MD, Principal Investigator — Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD), Hôpital l'Archet 2, 151 route Saint-Antoine de Ginestière 06202 Nice Cedex 3, France
Locations (1):
- Centre de Pharmacologie Clinique Appliquée à la Dermatologie (CPCAD), Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start date: 28-Jun-2012 Completion date: 15-Oct-2012
Pre-assignment Details: Prior to randomisation, the subjects entered a washout phase (if required) where antipsoriatic treatment and other relevant treatments had to be discontinued as defined by the exclusion criteria. Depending on prior use of disallowed treatments, the washout phase could last for up to 21 days.
Groups:
- Daivobet® Gel: Each of the 24 subjects participating in this exploratory trial received:
  * Daivobet® gel applied then removed after 10 minutes (+/- 2 minutes) : Once daily application, 3 weeks
  * Daivobet® gel vehicle applied for 24 hours (+/- 2 hours) : Once daily application, 3 weeks
  * Daivobet® gel applied then removed after 20 minutes (+/- 2 minutes) : Once daily application, 3 weeks
  * Daivobet® gel applied for 24 hours (+/- 2 hours) : Once daily application, 3 weeks
  The products were applied on 4 test sites of 2 cm according to random assignment to specific sites on one psoriasis plaque.
Period: Overall Study
Arm/Group | Daivobet® Gel
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daivobet® Gel
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Region of Enrollment [Number; unit: participants]
  France | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Clinical Score From Baseline to Day 22
Description: Investigator's rating of the clinical appearance of a psoriatic lesion. Maximum score is 9 (most severe); minimum score is 0 (least severe). The single items erythema, scaling, and infiltration (maximum score 3 each) are summed to obtain the Total Clincal Score
Time Frame: baseline to day 22
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Daivobet® Gel Applied Then Removed After 10 Minutes: Daivobet® gel applied then removed after 10 minutes (+/- 2 minutes) : Once daily application, 3 weeks
  The products were applied on 4 test sites of 2 cm according to random assignment to specific sites on one psoriasis plaque.
- Daivobet® Gel Applied Then Removed After 20 Minutes: - Daivobet® gel applied then removed after 20 minutes (+/- 2 minutes) : Once daily application, 3 weeks
  The products were applied on 4 test sites of 2 cm according to random assignment to specific sites on one psoriasis plaque.
- Daivobet® Gel Applied for 24 Hours: - Daivobet® gel applied for 24 hours (+/- 2 hours) : Once daily application, 3 weeks
  The products were applied on 4 test sites of 2 cm according to random assignment to specific sites on one psoriasis plaque.
- Daivobet® Gel Vehicle Applied for 24 Hours: Daivobet® gel vehicle applied for 24 hours (+/- 2 hours) : Once daily application, 3 weeks
  The products were applied on 4 test sites of 2 cm according to random assignment to specific sites on one psoriasis plaque.
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -3.6 (1.6) | -3.7 (2.0) | -4.9 (1.5) | -1.3 (0.9)

2. Secondary Outcome: Change in Total Clinical Score at Day 4 Compared to Baseline
Description: Investigator's rating of the clinical appearance of a psoriatic lesion. Maximum score is 9 (most severe); minimum score is 0 (least severe). The single items erythema, scaling, and infiltration (maximum score 3 each) are summed to obtain the Total Clinical Score.
Time Frame: Baseline to day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.5 (0.8) | -0.5 (0.6) | -0.4 (0.7) | -0.1 (0.5)

3. Secondary Outcome: Change in Total Clinical Score at Day 8 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline to day 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.5 (1.2) | -1.4 (1.4) | -1.6 (1.3) | -0.2 (0.9)

4. Secondary Outcome: Change in Total Clinical Score at Day 11 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline to day 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -2.3 (1.4) | -2.3 (1.4) | -3.0 (1.4) | -0.7 (1.0)

5. Secondary Outcome: Change in Total Clinical Score at Day 15 Compared to Baseline
Description: Investigator's rating of the clinical appearance of a psoriatic lesion. Maximum score is 9 (most severe); minimum score is 0 (least severe). The single items erythema, scaling, and infiltration (maximum score 3 each) are summed to obtain the Total Clinial Score.
Time Frame: Baseline to day 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -3.0 (1.3) | -2.8 (1.6) | -3.9 (1.5) | -0.9 (1.1)

6. Secondary Outcome: Change in Total Clinical Score at Day 18 Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline to day 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -3.4 (1.5) | -3.4 (1.6) | -4.3 (1.5) | -1.1 (1.0)

7. Secondary Outcome: Change From Baseline in Erythema at Day 4.
Description: Investigator's rating of the clinical appearance of erythema. Maximum score is 3 (most severe); minimum score is 0 (absent).
Time Frame: Baseline to day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.17 (0.32) | -0.23 (0.36) | -0.23 (0.36) | -0.06 (0.22)

8. Secondary Outcome: Change From Baseline in Erythema at Day 8.
Description: as for outcome 7
Time Frame: Baseline to day 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.54 (0.51) | -0.56 (0.50) | -0.67 (0.55) | -0.15 (0.35)

9. Secondary Outcome: Change From Baseline in Erythema at Day 11
Description: as for outcome 7
Time Frame: Baseline to day 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.79 (0.57) | -0.85 (0.52) | -1.06 (0.58) | -0.27 (0.36)

10. Secondary Outcome: Change From Baseline in Erythema at Day 15
Description: as for outcome 7
Time Frame: Baseline to day 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.00 (0.49) | -1.04 (0.62) | -1.29 (0.57) | -0.31 (0.48)

11. Secondary Outcome: Change From Baseline in Erythema at Day 18
Description: as for outcome 7
Time Frame: Baseline to day 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.04 (0.53) | -1.19 (0.53) | -1.42 (0.50) | -0.46 (0.41)

12. Secondary Outcome: Change From Baseline in Erythema at Day 22
Description: as for outcome 7
Time Frame: Baseline to day 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.17 (0.60) | -1.31 (0.66) | -1.56 (0.61) | -0.42 (0.41)

13. Secondary Outcome: Change From Baseline in Infiltration at Day 4
Description: Investigator's rating of the clinical appearance of infiltration. Maximum score is 3 (most severe); minimum score is 0 (absent).
Time Frame: Baseline to day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.10 (0.29) | -0.08 (0.28) | -0.10 (0.25) | 0.02 (0.10)

14. Secondary Outcome: Change From Baseline in Infiltration at Day 8
Description: as for outcome 13
Time Frame: Baseline to day 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.33 (0.38) | -0.33 (0.50) | -0.38 (0.47) | 0.00 (0.26)

15. Secondary Outcome: Change From Baseline in Infiltration at Day 11
Description: as for outcome 13
Time Frame: Baseline to day 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 2 | 24 | 24 | 24
units on a scale | -0.63 (0.52) | -0.60 (0.59) | -0.81 (0.53) | -0.08 (0.32)

16. Secondary Outcome: Change From Baseline in Infiltration at Day 15
Description: as for outcome 13
Time Frame: Baseline to day 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.81 (0.55) | -0.73 (0.63) | -1.19 (0.62) | -0.15 (0.28)

17. Secondary Outcome: Change From Baseline in Infiltration at Day 18
Description: as for outcome 13
Time Frame: Baseline to day 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.00 (0.59) | -0.98 (0.70) | -1.42 (0.65) | -0.17 (0.32)

18. Secondary Outcome: Change From Baseline in Infiltration at Day 22
Description: as for outcome 13
Time Frame: Baseline to day 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.08 (0.60) | -1.06 (0.74) | -1.60 (0.61) | -0.31 (0.32)

19. Secondary Outcome: Change From Baseline in Scaling at Day 4
Description: Investigator's rating of the clinical appearance of scaling. Maximum score is 3 (most severe); minimum score is 0 (absent).
Time Frame: Baseline to day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.19 (0.32) | -0.19 (0.29) | -0.10 (0.33) | -0.08 (0.35)

20. Secondary Outcome: Change From Baseline in Scaling at Day 8
Description: as for outcome 19
Time Frame: Baseline to day 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.60 (0.55) | -0.46 (0.57) | -0.56 (0.52) | -0.06 (0.45)

21. Secondary Outcome: Change From Baseline in Scaling at Day 11
Description: as for outcome 19
Time Frame: Baseline to day 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -0.90 (0.57) | -0.88 (0.45) | -1.08 (0.58) | -0.35 (0.50)

22. Secondary Outcome: Change From Baseline in Scaling at Day 15
Description: as for outcome 19
Time Frame: Baseline to day 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.15 (0.54) | -1.04 (0.55) | -1.40 (0.53) | -0.42 (0.55)

23. Secondary Outcome: Change From Baseline in Scaling at Day 18
Description: as for outcome 19
Time Frame: Baseline to day 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.35 (0.56) | -1.27 (0.61) | -1.50 (0.63) | -0.48 (0.45)

24. Secondary Outcome: Change From Baseline in Scaling at Day 22
Description: as for outcome 19
Time Frame: Baseline to day 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale | -1.31 (0.60) | -1.31 (0.70) | -1.71 (0.53) | -0.54 (0.41)

25. Secondary Outcome: Change in Lesion Thickness Measured by Ultrasound From Baseline to Day 22.
Time Frame: Baseline to day 22
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
millimeters | -0.61 (0.47) | -0.80 (0.57) | -0.90 (0.51) | -0.11 (0.26)

26. Secondary Outcome: Change in Skin Thickness - Echo-poor Band - Measured by Ultrasound From Baseline to Day 22
Time Frame: Baseline to day 22
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Daivobet® Gel Applied Then Removed After 10 Minutes | Daivobet® Gel Applied Then Removed After 20 Minutes | Daivobet® Gel Applied for 24 Hours | Daivobet® Gel Vehicle Applied for 24 Hours
Number analyzed (Participants) | 24 | 24 | 24 | 24
millimeters | -0.57 (0.35) | -0.54 (0.50) | -0.62 (0.33) | -0.06 (0.30)

ADVERSE EVENTS:
Arm/Group | Daivobet® Gel
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daivobet® Gel (N=24)
Nasopharyngititis (Infections and infestations) | 2
Headache (Nervous system disorders) | 2

LIMITATIONS AND CAVEATS:
In this small exploratory trial the subjects received all 4 investigational products on small dermal test sites.

Regarding Adverse Events, only local dermal reactions could be potentially attributed to a specific investigational product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is entitled to review and comment on publications prior to submission or presentation. Upon request of the sponsor, the investigator shall delay publication or presentation to allow for protection of the sponsors inventions and other intellectual property.